CLINICAL TRIAL: NCT01198106
Title: A Double-blind Randomized Placebo Controlled Comparison of Scopolamine With Cinnarizin for Prevention of Simulator Sickness
Brief Title: A Double-blind Comparison of Scopolamine With Cinnarizin for Prevention of Simulator Sickness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Amit Assa MD, IAF aeromedical center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 792-2008-IDF-CTIL
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Simulator Sickness
Keywords: simulator sickness; scopolamine; cinnarizine
MeSH Terms: interventions — Scopolamine; Cinnarizine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: scopolamine — 0.6 mg
  Other Names: kwells
Drug: cinnarizine — 50 mg
  Other Names: stonoron

SUMMARY:
BACKGROUND:flight simulator have become an important component in pilot training. However, they are known to be associated with motion sickness like symptoms defined as Simulator Sickness (SS). Prevention countermeasures against motion sickness have been studied extensively focusing on cholinergic blockers and antihistamines. Most comparataive studies emphasized the effectiveness of scopolamine over outher agents. Evidence, though, on prophylaxis against SS is sparse.

OBJECTIVE: to assess the effectiveness of oral scopolamine versus oral cinnarizine or placebo for SS prevention in helicopter pilots.

DESIGN: a prospective, placebo controlled double-blind.

SETTING: Israel Air Forse (IAF) Helicopter Aircaft vWeapon System Trainer.

PARTICIPANTS: IAF experienced helicopter pilots.

INTERVENTION: 0.6 mg oral scopolamine or 50 mg oral cinnarizine or placebo 1 hour before beginning of a 3 sortie simulator training

ELIGIBILITY:
Inclusion Criteria:

* age 21 to 50 years, qualified helicopter pilots
* history of average TS score in SSQ more than 7.48

Exclusion Criteria:

* known vestibular, visual or central nervous system pathology
* fever of more than 37.2 degrees
* any MS like symptom prior to simulator training
* any compromising acute health problem

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Finding more effective treatment to the motion sickness symptoms during and after simulator training. | 1 year
  To record a significant difference in motion sickness symptoms reduction during and after simulator training, after taking cinnarizine, scopolamine or placebo. We predict that scopolamine will prove to be more effective than cinnarizine with fewer side effects that can compromise pilot's performance during training.

CONTACTS AND LOCATIONS:
Locations (1):
- base 30 IAF, Yavné, Israel